CLINICAL TRIAL: NCT00276055
Title: Phase IB Study of Gemcitabine, Docetaxel and Bevacizumab in Patients With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0509C
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Sarcoma
Keywords: Soft Tissue Sarcoma; Phase I; Gemcitabine; Docetaxel; Bevacizumab; vascular endothelial growth factor
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): 1000mg/m2 gemcitabine
  Interventions: Drug: Gemcitabine, Docetaxel and Bevacizumab
- Cohort 2 (Experimental): 1250 mg/m2 gemcitabine
  Interventions: Drug: Gemcitabine, Docetaxel and Bevacizumab
- Cohort 3 (Experimental): 1500 mg/m2 gemcitabine
  Interventions: Drug: Gemcitabine, Docetaxel and Bevacizumab

INTERVENTIONS:
Drug: Gemcitabine, Docetaxel and Bevacizumab — During the treatment phase, pts. will receive the drug combination of gemcitabine, docetaxel, and bevacizumab every 2 weeks for a period of 4 weeks. This 4-week period is called a cycle of treatment. The treatment consists of receiving docetaxel IV over a 60-minute period and gemcitabine IV over a 30-minute period. Pts. will then receive bevacizumab IV over a 30-minute period. Pts. will receive this treatment once every 2 weeks. Pts. will receive at least 2 cycles of treatment unless you have progression of your disease or unmanageable side effects. As long as the size of pts.'s tumor stays the same or gets smaller, pts may continue receiving treatment
  Other Names: Taxotere; Gemzar; Avastin

SUMMARY:
1.1 To determine the recommended phase II dose for gemcitabine in combination with a fixed dose of docetaxel and bevacizumab.

1.2 To determine the efficacy of the combination of gemcitabine, docetaxel, and bevacizumab in patients with soft tissue sarcoma 1.3 To determine the toxicity profile of the combination of gemcitabine, docetaxel, and bevacizumab in patients with soft tissue sarcoma

DETAILED DESCRIPTION:
Because the combination of gemcitabine and docetaxel has shown impressive activity in soft tissue sarcoma, we hypothesize that the addition of an antiangiogenesis agent (bevacizumab) would enhance the anticancer activity, as shown in other tumor types.

ELIGIBILITY:
Inclusion criteria:

* All patients, 18 years of age or older, with chemotherapy naive soft tissue sarcoma are eligible if there is measurable disease Prior surgery or radiotherapy for the primary tumor is allowed but needs to have been completed at least 2 weeks from entry, and patient should have completely recovered from the procedures.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have a Zubrod performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of > 1,500 or cells/mm3 and platelet count >100,000/mm3 and absence of a regular red blood cell transfusion requirement.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.

Exclusion Criteria:

* Patients with symptomatic brain metastases are excluded from this study.
* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete and partial responses). | 4 years
  Tumor response is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). ORR is the sum of the percentages of patients achieving complete and partial responses

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (4):
- United States (4):
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico